CLINICAL TRIAL: NCT05685667
Title: Needless Laser Injector Versus Needle Injection for Antiaging Effect of Dermal Filler: A Randomized Split-face Comparison
Brief Title: Needless Laser Injector for Antiaging Effect of Dermal Filler
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jung-Won Shin, Associate Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIRAJET-KHIDI-2004
Record Dates: First submitted 2022-12-21; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Aging Problems
MeSH Terms: interventions — Needles

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser-induced microjet injector (Mirajet) (Experimental): The left/right assignment was sealed in a nontransparent envelop.
  Interventions: Device: needless laser injector (Mirajet)
- Needle injection (control) (Active Comparator): The left/right assignment was sealed in a nontransparent envelop.
  Interventions: Device: needle injection

INTERVENTIONS:
Device: needless laser injector (Mirajet) — Mirajet injection was performed 2-3 passes until a total of 2cc of diluted PLA/HA solution was completely injected to the one half of the face.
  Other Names: polylactic acid (PLA)/hyaluronic acid (HA) composite dermal filler
  Arms: Laser-induced microjet injector (Mirajet)
Device: needle injection — For traditional method of needle injection, intradermal injection using multi-puncture/micro-papule technique was used. A series of injections at 0.5-1 cm apart was performed on one half of the face so that a total of 2cc of diluted PLA/HA solution was injected.
  Other Names: polylactic acid (PLA)/hyaluronic acid (HA) composite dermal filler
  Arms: Needle injection (control)

SUMMARY:
The investigators aimed to evaluate the efficacy and safety of needless laser injector for antiaging effect of dermal filler.

DETAILED DESCRIPTION:
A 24-week prospective, single-center, assessor-blinded, randomized, split-face study was conducted to compare the clinical efficacy and safety of needless laser injector versus needle injection for anti-aging effect of dermal filler.

ELIGIBILITY:
Inclusion Criteria:

* patients who wanted to improve facial skin aging

Exclusion Criteria:

* a history of skin rejuvenation treatment (including filler, botulinum toxin, lasers, chemical peeling, and topical retinoid) within 6 month prior to the start of the study
* having a plan for skin rejuvenation treatment during the study
* current pregnancy or breastfeeding
* an allergy to polylactic acid (PLA) or hyaluronic acid (HA)
* uncontrolled medical diseases

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Skin hydration using a Corneometer® CM 825 | at 12 weeks after treatment

SECONDARY OUTCOMES:
Skin elasticity using a Cutometer® MPA 580 | at 12 weeks after treatment
Erythema index (EI) using a Mexameter® MX 18 (Courage & Khazaka) | at 12 weeks after treatment
Skin aging analyzed by three-dimensional photogrammetry | at 12 weeks after treatment
Patient's satisfaction score for antiaging effects | at 12 weeks after treatment
  from 1 (extremely dissatisfied) to 7 (extremely satisfied)
Patient's pain score during treatment | up to 24 weeks
  from 0 (none) to 10 (worst)
Adverse events related to the procedure | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jung Won Shin, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No